CLINICAL TRIAL: NCT00222703
Title: Enhancing Tobacco Abstinence Following Hospitalization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH); Eta Chapter, Sigma Theta Tau (Other); Pauline Thompson Clinical Research Award, Nursing Foundation of Pennsylvania (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1F31NR007343 (NIH)
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Last update posted 2005-09-22 (Estimated); Status verified 2005-09

CONDITIONS: Hospitalized Smokers; Chronic Diseases; Tobacco Use Disorder
Keywords: nicotine addiction; relapse; smoking; chronic disorders; randomized controlled trial; intervention
MeSH Terms: conditions — Chronic Disease; Tobacco Use Disorder; Recurrence; Smoking

INTERVENTIONS:
Behavioral: Smoking relapse prevention

SUMMARY:
The primary aim of this study is to examine the efficacy of a 12-week nurse-delivered relapse management intervention designed with conceptual underpinnings from Self-efficacy Theory to enhance smoking abstinence of hospitalized smokers following their hospital discharge. Specifically this study asks, does a 12-week Self-efficacy Theory driven relapse management intervention enhance smoking abstinence following hospitalization by increasing smoking abstinence point prevalence as measured by carbon monoxide validated self-reports of smoking, when compared to subjects receiving only enhanced usual care?

DETAILED DESCRIPTION:
A randomized controlled two-group design with an intent-to-treat approach for handling protocol deviations will be used to examine the primary aim of this project. The sample will consist of 80 consenting smokers prospectively recruited during hospitalization. Subjects will be randomly assigned by equal allocation to an intervention group or an enhanced usual only group. A baseline adaptive randomization procedure will adjust the random equal ratio of treatment assignment to maintain sampling balance of the groups for race (White/Black/Other), gender (male/female), and three comorbid categories (only tobacco related illnesses/ tobacco related and unrelated to tobacco illnesses/ unrelated to tobacco illnesses). All subjects will receive enhanced usual care, which will consist of receiving a supportive message to quit smoking and smoking cessation materials. Subjects assigned to the intervention group will receive 9 intervention sessions with a nurse aimed to enhance their self-efficacy in self-management of tobacco abstinence. These sessions will occur over 12 weeks following hospital discharge. All but the initial session will occur by telephone. Subjects will be asked to participate with follow-up activities 12 weeks and 24 weeks following their hospital discharge, which requires the measurement of exhaled carbon monoxide and the completion of questionnaires by self-administration and interview with study personnel. Subjects will exit from study following the 24-week follow-up.

ELIGIBILITY:
Inclusion Criteria:

* smoked one cigarette within 30 days of hospital admission
* admission to a medical/surgical patient care unit
* 18 years of age or older

Exclusion Criteria:

* diagnosis of cancer in a terminal state,
* under evaluation for organ transplantation or awaiting transplantation,
* cerebral vascular disorders,
* senile dementia,
* Alzheimer's disease,
* abstinence from smoking greater than one month,
* non-English speaking,
* lack of a home telephone,
* lack of a mailing address,
* lack of any ability to participate with self-care activities,
* and transfer to a rehabilitation hospital or nursing home following their hospital admission.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80
Dates: Start 2002-05; Study Completion 2005-03

PRIMARY OUTCOMES:
Self reported smoking status validated by exhaled CO

SECONDARY OUTCOMES:
Time to smoking lapse

CONTACTS AND LOCATIONS:
Overall Officials: Donna D Caruthers, PHD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States